CLINICAL TRIAL: NCT02429544
Title: Effects of a Group Residential Retreat on Cancer Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is unfunded and lack of resources
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2015-0011; NCI-2015-00717 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Stage IV breast cancer; Metastatic; Residential group programs; Questionnaires; Surveys; EEG; Computer testing; Saliva test; Study diary; Actigraph
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Surveys and Questionnaires; Electroencephalography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental Support Group (ESG) - Residential Program (Experimental): Participants attend a 7-day offsite, residential support program. On Day 5 of the program, participant joined by spouse or caregiver.
  Questionnaires completed at baseline visit, 1 month after baseline. EEG performed with simultaneous computer testing. Day after baseline visit, saliva collected for 3 days at different times to measure cortisol levels. For seven days after baseline visit, participants complete study diary describing sleeping habits. An actigraph also worn during this time to record physical activity and sleeping habits.
  Questionnaires and testing repeated 7 days after the residential program ends, and then again about 3 months later.
  Interventions: Behavioral: Residential Program; Behavioral: Questionnaires; Device: Electroencephalogram (EEG); Other: Saliva Testing; Behavioral: Study Diary plus Actigraph
- Standard Support Group (SSG) - Residential Program (Experimental): Participants attend a 7-day offsite, residential support program. On Day 5 of the program, participant joined by spouse or caregiver.
  Questionnaires completed at baseline visit, 1 month after baseline. EEG performed with simultaneous computer testing. Day after baseline visit, saliva collected for 3 days at different times to measure cortisol levels. For seven days after baseline visit, participants complete study diary describing sleeping habits. An actigraph also worn during this time to record physical activity and sleeping habits.
  Questionnaires and testing repeated 7 days after the residential program ends, and then again about 3 months later.
  Interventions: Behavioral: Residential Program; Behavioral: Questionnaires; Device: Electroencephalogram (EEG); Other: Saliva Testing; Behavioral: Study Diary plus Actigraph
- Standard of Care Group (SOC) - No Residential Program (Other): Questionnaires completed at baseline visit, 1 month after baseline. EEG performed with simultaneous computer testing. Day after baseline visit, saliva collected for 3 days at different times to measure cortisol levels. For seven days after baseline visit, participants complete study diary describing sleeping habits. An actigraph also worn during this time to record physical activity and sleeping habits.
  Questionnaires and testing repeated 7 days after the residential program ends, and then again about 3 months later.
  Interventions: Behavioral: Questionnaires; Device: Electroencephalogram (EEG); Other: Saliva Testing; Behavioral: Study Diary plus Actigraph

INTERVENTIONS:
Behavioral: Residential Program — Participants attend a 7-day offsite, residential support program. On Day 5 of the program, participant joined by spouse or caregiver.
  Other Names: Retreat
  Arms: Experimental Support Group (ESG) - Residential Program; Standard Support Group (SSG) - Residential Program
Behavioral: Questionnaires — Questionnaires completed about mood, sleep, fatigue, how participant has been feeling, and their general quality of life at baseline visit, 1 month after baseline, 7 days after residential program ends, and again about 3 months later.
  Other Names: Survey
Device: Electroencephalogram (EEG) — EEG performed at baseline with simultaneous computer testing consisting of 3 tests to check attention, short-term memory, and levels of emotions. EEG repeated 7 days after the residential program ends, and then again about 3 months later.
Other: Saliva Testing — Day after baseline visit, saliva collected for 3 days at different times to measure cortisol levels. Saliva testing repeated 7 days after the residential program ends, and then again about 3 months later.
Behavioral: Study Diary plus Actigraph — For seven days after baseline visit, participants complete study diary describing sleeping habits. An actigraph also worn during this time to record physical activity and sleeping habits.

SUMMARY:
The goal of this behavioral research study is to compare 2 different types of residential group programs to help researchers learn if and how well these groups may help to improve physical and emotional well-being in patients with stage IV breast cancer.

DETAILED DESCRIPTION:
Baseline Visit:

Signing this consent form does not mean that you will be able to take part in this study. The following baseline tests will help the doctor decide if you are eligible:

* You will complete 7 questionnaires about your mood, sleep, fatigue, how you have been feeling, and your general quality of life. The questionnaires should take about 60-80 minutes to complete.
* You will have an electroencephalogram (EEG) to check your brain's electrical activity. During the EEG, a snug cap with small electrodes will be placed on your head to measure the electrical patterns coming from the brain. This is like the way a doctor listens to your heart from the surface of your skin. During the EEG, you will complete 3 tests to check your attention, short-term memory, and levels of emotions on the computer. The study staff will discuss each test in more detail with you. The EEG and tests will take about 45-60 minutes total.
* If you have not had a computed tomography (CT) scan in the last 2 months, you will have one performed to check the status of the disease. If you have had one in the last 2 months, the results will be collected from your medical records.
* You will have an electrocardiogram (EKG) to check your heart function.
* Blood (about 6 tablespoons) will be drawn for tests to measure hormones and your immune system responses. You will need to fast (not eat or drink anything except water) for 12 hours before this blood draw. You will be provided with healthy snacks after your blood draw.

The day after your baseline visit, saliva will be collected to measure the level of cortisol (a type of stress hormone) in your body. These saliva samples will be collected 4 times each day for 3 days in a row. You will collect these samples at home when you first wake up, about 45 minutes later, about 10 hours after waking up, and then at bedtime. To collect each saliva sample, you will chew on a cotton ball for a few seconds and then put the cotton in a small plastic tube. You will write down the times you took these samples. You will mail these samples back to MD Anderson in postage-paid envelopes that will be provided to you. The tubes will also be provided at no cost to you. These saliva samples will be destroyed after being studied.

Every day for the next 7 days after your baseline visit, you will fill out a diary about your sleeping habits. You will also wear a special type of wrist watch for these 7 days. The watch will collect data about your physical activity and sleeping habits. After you have worn it for 7 days, you will mail the watch and the sleep diary back to MD Anderson in postage-paid envelopes that will be provided to you.

Extended Baseline:

You will be asked to complete and provide all the same measures again 1 month after the first baseline visit.

Study Groups:

If you are found to be eligible to take part in this study and you agree, you will be randomly assigned (as in the roll of dice) to 1 of 3 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group.

* If you are assigned to Groups 1 or 2, you will take part in 1 of 2 types of residential group programs.
* If you are assigned to Group 3, you will receive standard cancer care without any participation in a residential group program.

If you are assigned to Groups 1 or 2, neither you nor the study staff will know what kind of residential group program you are in.

Residential Support Program Sessions (Groups 1 and 2 only):

You will take part in a 7-day offsite, residential support program in groups of about 10 participants each. On Day 5 of the retreat, you will be joined by your spouse or caregiver.

During the 7 days, you will take part in group activities, learn relaxation skills, do different cognitive activities (for example, reading, watching movies, and having group discussions), and learn about mind-body connections. You will spend 7 days and 6 nights at the residential retreat. Activities at the retreat will last about 12 hours per day with breaks, group meals, and free time to rest in the morning, afternoon and evening, or as needed.

At least 1 week before the retreat, you will be given a detailed agenda and schedule of all activities that will occur during the retreat.

Follow-Up Sessions (All Groups):

You will complete the same tests/procedures that were performed at the baseline visit within 7 days after the residential program ends and then again about 3 months later. If you are in Group 3, you will complete the same tests/procedures on the same schedule.

Length of Participation:

Your participation on this study will be over after you complete the follow-up sessions.

Depending on which study group you were assigned to, you may be able to take part in a residential program that you did NOT previously take part in. The study chair or research staff will discuss this option with you.

This is an investigational study.

Up to 100 participants and their caregivers will take part in this multicenter study. Up to 74 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 50 and over initially diagnosed with breast cancer by histological tissue diagnosis in 2003 or later.
2. Currently Stage IV (metastatic) breast cancer on the basis of definitive imaging or biopsy with stable disease (scans within the past 2 months).
3. ECOG (Eastern Cooperative Group) Performance Score of 0 or 1.
4. Able to participate occasionally in mildly strenuous physical effort.
5. Able to read, speak, and write in English or ability to provide consent or understand questionnaires.
6. Able to be accompanied by their spouse or significant other partner/friend (spouse, significant other, partner, or friend.
7. Able to travel to the retreat site.
8. Must be right handed.
9. Patients must have had a contrast-enhanced computerized tomographic (CT) scan of the chest and abdomen within 2 months of study entry and be willing to have a follow up scan within 2 months of the completion of the retreat.
10. (CAREGIVERS ONLY) Must be primary caregiver of the patient.
11. (CAREGIVERS ONLY) Able to read, speak, and write in English.
12. (CAREGIVERS ONLY) Able to attend the last two days of the retreat with patient.

Exclusion Criteria:

1. Significant co-morbidities (e.g., diabetes, cardiac disease, or other condition that in the opinion of the primary physician or investigators would limit participation in the intervention groups) that would preclude study participation.
2. Evidence of disease progression that would necessitate a treatment in the next 2 weeks.
3. Need for intravenous therapy more frequently than every 3 weeks or inability to time intravenous therapy treatment before and after the study.
4. Currently in treatment for a major psychiatric disorder
5. Clinical history of severe psychiatric disorders.
6. Currently receiving chemotherapy.
7. (CAREGIVERS ONLY) Must be an adult (>=18 years old).

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Compliance in Residential Retreat Program | 3 months
  Participant compliance with assessments monitored as well as participation in all aspects of the intervention program. Intervention deemed feasible if ≥ 60% of enrolled couples complete all assessments and attend the assigned retreat.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PHD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org